CLINICAL TRIAL: NCT05606965
Title: Phase 2, Open-Label Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1010 and Comparator Seasonal Influenza Vaccines in Healthy Adults
Brief Title: A Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1010 in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: mRNA-CRID-003
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Influenza
Keywords: mRNA-1010; Influenza Vaccine; Moderna
MeSH Terms: conditions — Influenza, Human | interventions — mRNA-1010 influenza vaccine; fluarix; fluad vaccine; Influenza Vaccines; mRNA-1345 respiratory syncytial virus vaccine

STUDY DESIGN:
Intervention Model Description: The study design for Part A and Prt C is randomized and Part B is non-randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Parts A and B - Arm 1: mRNA-1010 (Age Group 18-50 years) (Experimental): Participants will receive a single dose of mRNA-1010 by intramuscular (IM) injection on Day 1.
  Interventions: Biological: mRNA-1010
- Parts A and B - Arm 2: Egg-based Quadrivalent Influenza Vaccine (Age Group 18-50 years) (Active Comparator): Participants will receive a single dose of egg-based quadrivalent influenza vaccine by IM injection on Day 1.
  Interventions: Biological: Egg-based Quadrivalent Influenza Vaccine
- Parts A and B - Arm 3: Adjuvanted Quadrivalent Influenza Vaccine (Age Group 65-80 years) (Active Comparator): Participants will receive a single dose of adjuvanted quadrivalent influenza vaccine by IM injection on Day 1.
  Interventions: Biological: Adjuvanted Quadrivalent Influenza Vaccine
- Parts A and B - Arm 4: Inactivated Influenza Vaccine (Age Group 65-80 years) (Active Comparator): Participants will receive a single dose of inactivated influenza vaccine by IM injection on Day 1.
  Interventions: Biological: Inactivated Influenza Vaccine
- Parts A and B - Arm 5: mRNA-1010 (Age Group 65-80 years) (Experimental): Participants will receive a single dose of mRNA-1010 by IM injection on Day 1.
  Interventions: Biological: mRNA-1010
- Part C - Arm 1: mRNA-1010 and mRNA-1345 (Age Group 18-50 years) (Experimental): Participants will receive one dose of mRNA-1010 concomitantly injected with one dose of mRNA-1345 in the contralateral arm at Day 1.
  Interventions: Biological: mRNA-1010; Biological: mRNA-1345
- Part C - Arm 2: mRNA-1010 and mRNA-1345 (Age Group 18-50 years) (Experimental): Participants will receive one dose of mRNA-1010 at Day 1 followed by one dose of mRNA-1345 in the contralateral arm at Day 29.
  Interventions: Biological: mRNA-1010; Biological: mRNA-1345
- Part C - Arm 3: mRNA-1045 (Age Group 18-50 years) (Experimental): Participants will receive a single dose of mRNA-1045 by IM injection on Day 1.
  Interventions: Biological: mRNA-1045

INTERVENTIONS:
Biological: mRNA-1010 — Sterile liquid for injection
  Arms: Part C - Arm 1: mRNA-1010 and mRNA-1345 (Age Group 18-50 years); Part C - Arm 2: mRNA-1010 and mRNA-1345 (Age Group 18-50 years); Parts A and B - Arm 1: mRNA-1010 (Age Group 18-50 years); Parts A and B - Arm 5: mRNA-1010 (Age Group 65-80 years)
Biological: Egg-based Quadrivalent Influenza Vaccine — Sterile suspension for injection
  Other Names: Fluarix®
  Arms: Parts A and B - Arm 2: Egg-based Quadrivalent Influenza Vaccine (Age Group 18-50 years)
Biological: Adjuvanted Quadrivalent Influenza Vaccine — Sterile injectable emulsion
  Other Names: Fluad®
  Arms: Parts A and B - Arm 3: Adjuvanted Quadrivalent Influenza Vaccine (Age Group 65-80 years)
Biological: Inactivated Influenza Vaccine — Sterile suspension for injection
  Other Names: Fluzone®
  Arms: Parts A and B - Arm 4: Inactivated Influenza Vaccine (Age Group 65-80 years)
Biological: mRNA-1345 — Sterile liquid for injection
  Arms: Part C - Arm 1: mRNA-1010 and mRNA-1345 (Age Group 18-50 years); Part C - Arm 2: mRNA-1010 and mRNA-1345 (Age Group 18-50 years)
Biological: mRNA-1045 — Sterile liquid for injection
  Arms: Part C - Arm 3: mRNA-1045 (Age Group 18-50 years)

SUMMARY:
The main purpose of the study is to evaluate the safety, reactogenicity, and the humoral immunogenicity of mRNA-1010 and comparator influenza vaccines against homologous influenza A and B strains at Day 29.

DETAILED DESCRIPTION:
The study consists of 3 parts. Part A of the study was conducted for the 2022-23 influenza season. Part B of the study was conducted in 2023-24 influenza season. Part C of the study will be conducted in 2024-25 influenza season.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-50 years (Study Parts A, B, and C) and 65-80 years (Study Parts A and B only) of age at the time of consent (Screening Visit).
* Part A only: Body mass index (BMI) of 18 kilograms (kg)/meter (m)^2 to < 40 kg/m^2 at the Screening Visit. There will be no BMI requirement for inclusion in Part B and Part C.
* A person of childbearing potential (POCBP): has a negative highly sensitive pregnancy test at the Screening Visit and before each administration of study intervention; must use a contraceptive method that is highly effective from at least 28 days prior to Day 1 (Baseline) to at least 3 months after the last study intervention; and is not currently pregnant or breastfeeding.

Exclusion Criteria:

* Acutely ill or febrile (temperature ≥ 38.0°Celsius (C)/100.4° Fahrenheit (F) hours before or at the D1 vaccination visit. Participants meeting this criterion may be rescheduled within the 28-day screening window.
* Any medical, psychiatric, or occupational condition, including reported history of substance abuse, that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* Reported history of congenital or acquired immunodeficiency, immunocompromizing or immunosuppressive condition, asplenia, or history of recurrent severe infections. Certain immune-mediated conditions that are stable and well-controlled (for example, Hashimoto's thyroid disease) or that do not require systemic immunosuppressive therapy may be permitted at the discretion of the Investigator.
* Dermatologic conditions that could affect local solicited AR assessments (tattoos, psoriatic patches or vitiligo affecting skin over the deltoid injection site area).
* Has received systemic immunosuppressants (for glucocorticoids ≥ 10 mg/day of prednisone or equivalent) for > 14 days in total within 180 days before vaccination visit (D1) or is anticipating the need for systemic immunosuppressive treatment at any time during participation in the study (including intra-articular steroid injections). Inhaled, nasal, and topical steroids are allowed.
* Has received systemic immunoglobulins or long-acting biological therapies that may suppress or alter immune responses (for example, Infliximab®) or blood products within 90 days before the vaccination visit or plans to receive them during the study.
* Has a history of anaphylaxis or severe hypersensitivity reaction after receipt of any mRNA or influenza vaccines or any components of the mRNA or influenza vaccines, including egg protein.

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Parts A, B, and C: Number of Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs) | Up to Day 7 (7 days after vaccination)
Parts A, B, and C: Number of Unsolicited Adverse Events (AEs) | Up to Day 28 (28 days after vaccination)
Parts A, B, and C: Number of Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs), Medically Attended Adverse Events (MAAEs), and AEs Leading to Discontinuation | Day 1 through Day 181
Parts A, B, and C: Geometric Mean Titer (GMT) of Anti-Hemagglutinin (HA) Antibodies at Day 29, as Measured by Hemagglutinin Inhibition (HAI) Assay | Day 29
Part C: GMT of Anti-Respiratory Syncytial Virus (RSV) Antibodies at Day 29, as Measured by Microneutralization Assay for RSV A and B | Day 29
Parts A, B, and C: Geometric Mean Fold Rise (GMFR) of Anti-HA Antibodies at Day 29, as Measured by HAI Assay | Baseline, Day 29
Part C: GMFR of Anti-RSV Antibodies at Day 29, as Measured by Microneutralization Assay | Baseline, Day 29
Parts A, B, and C: Percentage of Participants with Seroresponse at Day 29, as Measured by HAI Assay | Day 29
  Seroresponse is defined as a Day 29 titer > 1:40 if baseline is < 1:10 or a minimum 4-fold rise if baseline is >1:10 in anti-HA antibodies measured by HAI assay.
Part C: Percentage of Participants with Seroresponse at Day 29, as Measured by RSV Neutralization Assay | Day 29
  Seroresponse is defined as post-baseline titer ≥4-fold if baseline is ≥LLOQ or ≥4×LLOQ if baseline titer is <LLOQ in neutralizing antibody titers measured by RSV neutralization assay, at Day 29.

SECONDARY OUTCOMES:
Parts A and B: GMT of Anti-HA Antibodies at Days 121 and 181, as Measured by HAI Assay or Microneutralization Assay | Days 121 and 181
Part C: GMT of Anti-HA Antibodies at Days 57, 121, and 181, as Measured by HAI Assay or Microneutralization Assay | Days 57, 121, and 181
Parts A and B: GMFR of Anti-HA Antibodies at Days 121 and 181, as Measured by HAI Assay or MN Assay | Baseline, Days 121 and 181
Part C: GMFR of Anti-HA Antibodies at Days 57, 121, and 181, as Measured by HAI Assay or MN Assay | Baseline, Days 57, 121, and 181
Part C: Percentage of Participants with Seroresponse at Days 57, 121, and 181, as Measured by HAI Assay | Days 57, 121, and 181
  Seroresponse is defined as a Day 57, 121, or 181 titer > 1:40 if baseline is < 1:10 or a minimum 4-fold rise if baseline is >1:10 in anti-HA antibodies measured by HAI assay.
Part C: Percentage of Participants with Seroresponse at Days 57, 121, and 181, as Measured by RSV Neutralization Assay | Days 57, 121, and 181
  Seroresponse is defined as post-baseline titer ≥4-fold if baseline is ≥LLOQ or ≥4×LLOQ if baseline titer is <LLOQ in neutralizing antibody titers measured by RSV neutralization assay, at Days 57, 121, or 181.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States